CLINICAL TRIAL: NCT03541785
Title: Use of NGAL to Optimize Fluid Dosing, CRRT Initiation and Discontinuation in Critically Ill Children With Acute Kidney Injury
Brief Title: Use of NGAL for Fluid Dosing and CRRT Initiation in Pediatric AKI
Acronym: Taking Focus 2
Status: Enrolling by invitation | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: CIN001 - Taking Focus 2; 2P50DK096418-06 (NIH)
Record Dates: First submitted 2018-05-16; First posted 2018-05-31 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Injury; Renal Replacement Therapy; Pediatric Intensive Care Units
Keywords: NGAL; Renal Angina Index
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study follows a group of patients admitted to the PICU who are identified as being at risk for developing acute kidney injury. The investigators will use risk-stratification, biomarker testing, and a functional assessment to predict patients who will become fluid overloaded and develop acute kidney injury.

DETAILED DESCRIPTION:
In the pediatric population, acute kidney injury (AKI) is commonly observed in critically ill patients. At this time, there are no standardized care pathways that begin at identifying patients at risk for developing AKI and progress through to early recognition and treatment. Through previous work, the investigators have developed, tested, and integrated an AKI risk-stratification/clinical recognition tool (RAI) and a urine biomarker (NGAL) to try to identify patients at risk vs. not at-risk for developing AKI. However, these factors alone have yet to be integrated into clinical decision support to optimize AKI therapies and patient outcomes. The furosemide stress test (FST), previously described in adults, may be a good predictor for the patients who need acute dialysis for AKI versus those that can be managed medically.

Through this study, the investigators will be following a cohort of patients admitted to the PICU who are identified as being at risk for developing AKI through RAI and NGAL results. The aim is to standardize the FST in this population, as well as determine the accuracy of the RAI-NGAL-FST clinical decision tool in predicting patients who become fluid overloaded and develop AKI.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Pediatric Intensive Care Unit (PICU)
* Renal Angina Index (RAI) greater than or equal to 8
* Urine NGAL greater than or equal to 150 ng/mL
* Indwelling urinary catheter

Exclusion Criteria:

* Evidence of volume depletion
* Baseline Chronic Kidney Disease (CKD) Stage IV or V (estimated GFR <60 mL/min/1.73m2)
* History of kidney transplantation
* Active DNR order or clinical team is not committed to escalating medical care
* Known history of allergic reaction to furosemide (only for FST)

Ages: 3 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All critically ill patients admitted to the PICU at Cincinnati Children's Hospital Medical Center at risk for developing Acute Kidney Injury
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Decision Support Success (CDS) | 48 hours of PICU admission
  Time to complete risk stratification (RAI), biomarker testing (NGAL), and functional kidney assessment (FST) is less than 48 hours

SECONDARY OUTCOMES:
Furosemide Stress Test (FST) Standardization | 12 months
  Validate FST in critically ill pediatric patients, with a standard dose and urinary response

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Goldstein, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided